CLINICAL TRIAL: NCT04109118
Title: Distress Tolerance and Benzodiazepine Discontinuation in Opioid Agonist Therapy, Phase 2
Brief Title: Benzodiazepine Discontinuation in Opioid Agonist Therapy
Acronym: BZD-OAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-38981; 1K23DA044321-01 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Substance Use Disorders
Keywords: Opioid agonist therapy; Benzodiazepine; Distress tolerance; Distress Tolerance - Benzodiazepine Discontinuation (DT-BD); Relaxation Therapy (RT)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Benzodiazepines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Distress Tolerance - Benzodiazepine Discontinuation (DT-BD) (Other): This psychosocial treatment intervention uses a combination of interoceptive exposure therapy and elements of acceptance and commitment therapy (ACT) and psychoeducation about benzodiazepine use in OAT.
  Of note, this is a pilot trial for feasibility and acceptability. There is no randomization and we are not comparing arms.
  Interventions: Behavioral: Distress Tolerance - Benzodiazepine Discontinuation (DT-BD); Drug: BZD discontinuation protocol

INTERVENTIONS:
Behavioral: Distress Tolerance - Benzodiazepine Discontinuation (DT-BD) — Distress Tolerance - Benzodiazepine Discontinuation (DT-BD) is a psychosocial intervention. It is paired with a benzodiazepine taper. The aim of the psychosocial intervention is to improve individuals' ability to tolerate distress in order to assist benzodiazepine discontinuation in patients treated with OAT. There will be 5 sessions between therapist and participant prior to the start of the benzodiazepine taper. The taper for both the intervention and control conditions occurs over 9 weeks and involves weekly meetings with a benzodiazepine prescriber during which a gradual benzodiazepine dose reduction will take place. The DT-BD intervention combines elements of existing psychosocial interventions. Specifically, interoceptive exposure techniques will be paired with elements of acceptance and commitment therapy (ACT) and relapse prevention (RP).
Drug: BZD discontinuation protocol — All participants will undergo BZD discontinuation. Once the starting BZD dose is determined by prescription monitoring and/or self-report, we will maintain participants on this dose until the start of the BZD taper. Participants will see a study physician weekly to receive their BZD medication for the week until the taper is completed. BZD discontinuation in this study will consist of a gradual BZD taper in dose over 9 weeks. The taper will be flexible in that the study physician will utilize clinical judgement to lengthen the taper if necessary, depending on the severity of the participant's withdrawal symptoms. Anchor points will be set (33% reduction in dose after 2 weeks, 50% mid-treatment, 100% by week 8) to emphasize the time-limited nature of the taper.
  Other Names: Benzodiazepine

SUMMARY:
The proposed study is a clinical trial, designed to pilot test a Distress Tolerance-Benzodiazepine Discontinuation (DT-BD) intervention for patients on opioid agonist therapy who currently use benzodiazepines. The DT-BD intervention is an adjunctive psychosocial intervention in people seeking to discontinue (BZD) use. The goal of the study is to assess the applicability and feasibility of this intervention through treatment retention and qualitative interviews with four participants who are receiving opioid agonist treatment and who regularly use BZDs.

DETAILED DESCRIPTION:
This study pilots a 13-week psychosocial intervention paired with a benzodiazepine taper with the aim of assisting individuals receiving OAT discontinue benzodiazepine use. All participants will receive the same benzodiazepine (BZD) discontinuation protocol. The Distress Tolerance-Benzodiazepine Discontinuation (DT-BD) intervention consists of 14 study visits: the first visit consists of the baseline assessment and the first therapy visits, 4 subsequent weekly therapy visits, then a 9-week BZD taper. Some participants may be prescribed non-benzodiazepine medications to treat the underlying conditions for which they were using BZDs [e.g. selective serotonin reuptake inhibitors (SSRI) for anxiety or hypnotics for insomnia]. Data collection will occur starting at the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Receiving OAT (methadone or buprenorphine) confirmed by toxicology testing for at least 90 days and on a steady dose for 2 consecutive weeks
3. Regular BZD use defined by BZD use 3 or more times per week in past month by self-report and positive urine screen at time of recruitment
4. Provides permission to contact current BZD prescriber if being prescribed BZDs
5. Speaks English
6. Wants to discontinue BZD use

Exclusion Criteria:

1. Pregnant, confirmed by urine pregnancy test
2. Cognitive impairment, as indicated by a score of < 23 on the Mini Mental Status Exam
3. Any past month illicit opioid, barbiturate, z-drug, cocaine, unprescribed amphetamine, or synthetic cannabinoid use determined by self-report or urine drug test
4. Receiving ongoing psychosocial treatment for BZD use disorder
5. Uncontrolled seizure disorder (i.e. seizure in prior 90 days), or past BZD withdrawal seizure
6. Current suicidality or homicidality
7. Current psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Woo Park, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began in March 2021. Potential participants identified by the study PI were given study information and PI obtained verbal consent from patients to have study staff call to invite them to participate over the phone. Interested potential participants were asked to complete a brief screening interview using the study screening script that involved asking questions based on the inclusion and exclusion criteria.
Groups:
- Distress Tolerance - Benzodiazepine Discontinuation (DT-BD): This is a pilot clinical trial of the DT-BD intervention. The study population will consist of outpatients receiving OAT for opioid use disorder who are also using BZDs regularly. All participants will receive the same BZD discontinuation protocol.
  DT-BD is paired with a benzodiazepine taper. The aim of the psychosocial intervention is to improve individuals' ability to tolerate distress in order to assist BZD discontinuation in patients treated with OAT. There will be 5 sessions between therapist and participant prior to the start of the BZD taper. The taper occurs over 9 weeks and involves weekly meetings with a BZD prescriber during which a gradual BZD dose reduction will take place.
  Once the starting BZD dose is determined by prescription monitoring and/or self-report, we will maintain participants on this dose until the start of the BZD taper. Participants will see a study physician weekly to receive their BZD medication for the week until the taper is completed. BZD discontinuation in this study will consist of a gradual BZD taper in dose over 9 weeks. The taper will be flexible in that the study physician will utilize clinical judgement to lengthen the taper if necessary, depending on the severity of the participant's withdrawal symptoms. Anchor points will be set (33% reduction in dose after 2 weeks, 50% mid-treatment, 100% by week 8) to emphasize the time-limited nature of the taper.
Period: Overall Study
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Started | 4
Completed | 1
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Self-report on drug use in the past 30 days [Count of Participants; unit: Participants]
  Used drug | 0
  Did not use drug | 4
Urine drug screen [Count of Participants; unit: Participants]
  Positive | 0
  Negative | 4
Psychiatric diagnostic interview [Count of Participants; unit: Participants]
  Panic Disorder Current + substance use disorder | 1
  Obsessive Compulsive Disorder + Major depressive disorder | 1
  Major Depressive Disorder | 1
  Alcohol use disorder +Bipolar I Disorder (past): depressed | 1
Highest level of education [Count of Participants; unit: Participants]
  8th grade or less | 0
  8-12th grade, no diploma | 0
  High school graduate or GED complete | 3
  Completed a vocational, trade, or business school program | 1
  Some college, no degree | 0
  Associate Degree | 0
  Bachelor's Degree | 0
  Master's Degree | 0
  Doctorate Degree | 0
Sexual orientation [Count of Participants; unit: Participants]
  Heterosexual | 3
  Homosexual | 0
  Bisexual | 1
  Other | 0
Do you have children [Count of Participants; unit: Participants]
  Yes | 2
  No | 2
Marital Status [Count of Participants; unit: Participants]
  Married | 0
  Not married, but living with a partner | 1
  Never married | 2
  Divorced | 1
Ever been prescribed a BZD by a professional [Count of Participants; unit: Participants]
  Yes | 4
  No | 0
Reason for being prescribed BZD [Count of Participants; unit: Participants]
  Anxiety | 3
  Other Psychiatric Disorder | 1
  Depression | 0
  Sleep | 0
  Pain | 0
Currently prescribed BZD [Count of Participants; unit: Participants]
  Yes | 3
  No | 1
Ever used BZD without a prescription [Count of Participants; unit: Participants]
  Yes | 2
  No | 2
First source of nonmedical BZD [Count of Participants; unit: Participants]
  Given by acquaintance | 1
  Given by family member | 1
  Not applicable | 2
Reason for using nonmedical BZD [Count of Participants; unit: Participants]
  To get high/for eurphoria | 1
  Help with panic attack | 1
  Not applicable | 2
Ever used nonmedical BZD at least 3 times a week [Count of Participants; unit: Participants]
  Yes | 1
  No | 1
  N/A | 2
Used nonmedical BZD in the past 12 months [Count of Participants; unit: Participants]
  Yes | 1
  No | 1
  N/A | 2
Frequency of using nonmedical benzodiazepine to relax [Count of Participants; unit: Participants]
  often | 1
  N/A | 3
Breath holding exercise (in seconds) [Mean (Standard Deviation); unit: seconds] | 54.5 (39.5)
Pittsburgh Sleep Quality Index rate sleep quality [Count of Participants; unit: Participants] — Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), a 9 item self report instrument, designed to measure quality and patterns of sleep from very good to very bad.
  Participants
    Very Good | 1
    Fairly good | 1
    Fairly bad | 0
    Very bad | 2
How helpful were the information and skill from this session? [Count of Participants; unit: Participants]
  not at all helfpful | 0
  A little helpful | 0
  Somewhat helpful | 0
  Very helpful | 1
  Extremely helpful | 3
How well did you understand the information and skills presented in the session? [Count of Participants; unit: Participants]
  did not undrestand | 0
  Understood a little | 0
  Understood some | 0
  Understood very well | 1
  Understood extremely well | 3
Distress Intolerance Index [Mean (Standard Deviation); unit: seconds] — Distress tolerance will be assessed with the computerized Mirror Tracing Persistence Task (MTPT-C). It is a computerized version of the original Mirror Tracing Persistence Task in which trace multiple progressively difficult polygons, with participants free to terminate at any point. Distress tolerance is measured by the latency in seconds to task termination.
  seconds | 16 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Participant Acceptability of the Interventions
Description: Number of participants who rated the intervention as acceptable, this was assessed by conducting an in-depth exit interview with the participant once they complete the entire 13-week study.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Thought that the program was acceptable and feasible | 1
  Thought that the program was not acceptable and feasible | 0

2. Primary Outcome: Number of Participants Who Rates the Intervention as Feasible
Description: Feasibility of intervention will be measured through the number of participants recruited and enrolled in the study, number of participants who started the BZD taper, and completed assessment tools.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Completion of Intervention
Description: Completion of intervention will be measured through participant attendance of weekly sessions. Participants must attend all 13 sessions (Baseline, 3 weekly therapy sessions prior to taper, and 8 week BZD taper urine/drug screens). Participants, who miss a study visit, will be considered discontinued from the study if study staff are unable to get in contact with them 7 days after their missed study visit.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: BZD Use Based on Self-report
Description: Timeline follow-back will be measured using the 30-day Timeline Followback (TLFB), adapted for BZD use. The Timeline Followback (TLFB) is a clinical and research method to obtain quantitative estimates of drug or alcohol use, and change over time. Participants will be asked to retrospectively estimate their BZD use 7 days prior to study visit. We will also monitor BZD use on a daily basis with a mobile phone application.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Used Drugs | 0
  Did not use drugs | 1

5. Secondary Outcome: Illicit Drug Use Based on Urine Drug Tests
Description: Illicit drug use urine tests will screen for amphetamines, benzodiazepines, opiates, oxycodone, fentanyl, cocaine, barbiturates, and methadone. Plus: liquid chromatography-mass spectrometry for clonazepam and lorazepam, and fentanyl if fentanyl test (immunoassay) is positive.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Used drugs | 0
  Did not use drugs | 1

6. Secondary Outcome: Alcohol Use Based on Urine Drug Tests
Description: Urine drug tests will include a ethyl glucuronide (EtG) test to detect the presence in the urine of ethyl glucuronide.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Did not use alcohol | 1
  Used alcohol | 0

7. Secondary Outcome: Alcohol Use Based on Self-report
Description: Timeline follow-back will be measured using the 30-day Timeline Followback (TLFB). The Timeline Followback (TLFB) is a clinical and research method to obtain quantitative estimates of drug or alcohol use, and change over time. Participants will be asked to retrospectively estimate their alcohol use 7 days prior to study visit. The alcohol adaption includes estimates of 1 standard drink in terms of beer, wine, and hard liquor. We will also monitor alcohol use on a daily basis with a mobile phone application.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Used alcohol | 0
  Did not use alcohol | 1

8. Secondary Outcome: BZD Withdrawal Symptoms
Description: BZD withdrawal symptoms will be measured using the Clinical Institute Withdrawal Assessment-Benzodiazepines (CIWA-B). The CIWA-B is a 20 item instrument, to assess severity of benzodiazepine withdrawal, including nausea and vomiting, anxiety, tremor, sweating, auditory disturbances, visual disturbances, tactile disturbances, headache, agitation, and clouding of sensorium. Scores range from 0 to 80, with 1-20 mild withdrawal, 21-40 moderate withdrawal, 41-60 severe withdrawal, and 61-80 very severe withdrawal.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  mild withdrawal (total score 1-20) | 1
  severe withdrawal (Total score 21-40) | 0
  very severe withdrawal (Total score 41-80) | 0

9. Secondary Outcome: Anxiety Symptoms
Description: The Overall Anxiety Severity and Impairment Scale (OASIS) is a 5-item self-report measure that can be used to assess severity and impairment associated with any anxiety disorder or multiple anxiety disorders.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  no severity and impairment associated with any anxiety disorder | 1
  severity and impairment associated with any anxiety disorder | 0

10. Secondary Outcome: Depressive Symptoms
Description: The Patient Health Questionnaire (PHQ)-9 is the major depressive disorder (MDD) module of the full PHQ.
  It is used to diagnose depression and grade severity of symptoms in general medical and mental health settings.
  Scores each of the 9 DSM criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  no depression | 1
  depression present | 0

11. Secondary Outcome: Sleep Quality
Description: Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), a 9 item self report instrument, designed to measure quality and patterns of sleep from very good to very bad. Sleep quality will also be measured on a daily basis with a mobile phone application. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  total score above 5 | 1
  total score below 5 | 0

12. Secondary Outcome: Inability to Tolerate Negative States
Description: The Distress Intolerance (DI) Index will be used to assess Inability to tolerate negative states.The index is a 10 item self-report measure designed to assess the inability to tolerate negative states. Items are rated from 0 (very little) to 4 (very much) and are summed for a total score, with higher scores indicating greater DI.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
score on a scale | 3 (0)

13. Secondary Outcome: Inflexibility or Experiential Avoidance
Description: The Acceptance and Action Questionnaire-II will be used to measure inflexibility or experiential avoidance. It is a 7 item self-report measure of psychological inflexibility or experiential avoidance. Each of the 7 items can be rated on a scale of 1 (never true) to 7 (always true) so scores can range from 7 to 49. Higher scores equal greater levels of psychological inflexibility.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
score on a scale | 3 (0)

14. Secondary Outcome: Fear of Anxiety Symptoms
Description: Fear of anxiety symptoms will be assessed by the Anxiety Sensitivity Index. It is a 16 item scale with each item rated on a five-point Likert scale ranging from 0 (very little) to 4 (very much). Scores can range from 0 to 64. Higher scores reflect greater fear of anxiety symptoms.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
score on a scale | 10 (0)

15. Secondary Outcome: Number of Participants Assessed for Distress Tolerance
Description: Distress tolerance will be assessed with the computerized Mirror Tracing Persistence Task (MTPT-C). It is a computerized version of the original Mirror Tracing Persistence Task in which trace multiple progressively difficult polygons, with participants free to terminate at any point. Distress tolerance is measured by the latency in seconds to task termination.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants
  Mirror Tracing Complete | 1
  Mirror Tracing Incomplete | 0

16. Secondary Outcome: Number of Participants Assessed for Motivations to Use BZD
Description: BZD motivations will be measured using the 12 item BZD Motivation Scale, a self report questionnaire. The questionnaire uses a 4 point Likert scale to assess participant motivations for using BZD, such as managing pain, insomnia, anxiety, and increase high of other illicit drugs.
Time Frame: 13 weeks
Population: 3 out of the 4 participants were lost to follow-up prior to the collection of this primary outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 13 weeks
Groups:
- Distress Tolerance - Benzodiazepine Discontinuation (DT-BD): The study population will consist of outpatients receiving OAT for opioid use disorder who are also using BZDs regularly. All participants will receive the same BZD discontinuation protocol.
Arm/Group | Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
There was an intended sample of four participants, and only one out of the four participants completed the whole 13-week study. This is due to the barrier of coming in-person for their weekly appointment during the peak of COVID-19 pandemic when the vaccines were just becoming available to the public.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT04109118/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04109118/ICF_000.pdf